CLINICAL TRIAL: NCT00181909
Title: Efficacy of Proactive Telephone Counseling for Pregnant Smokers Enrolled in a Managed Care Organization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000-P-002438
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2005-09

CONDITIONS: Pregnancy; Smoking Cessation
Keywords: Pregnancy; Smoking cessation
MeSH Terms: conditions — Smoking Cessation

INTERVENTIONS:
Behavioral: Smoking cessation counseling delivered by telephone

SUMMARY:
The principal objective is to test whether offering pregnant smokers a proactive telephone counseling program throughout pregnancy and for 2 months postpartum increases the rate of smoking cessation at end of pregnancy and 3 months postpartum, compared to a "best practice" control condition.

DETAILED DESCRIPTION:
A randomized controlled trial compared the efficacy of a proactive pregnancy-tailored telephone-delivered smoking cessation counseling program with a "best practice" brief counseling control condition among pregnant women referred by prenatal care providers and a managed care plan in Massachusetts. Intervention group patients received up to 105 min of cognitive-behavioral counseling delivered in a motivational interviewing style by trained counselors throughout pregnancy and for 2 months postpartum. Control group patients received 5 minutes of brief counseling at 1 telephone call. All participants were mailed written self-help smoking cessation material tailored to pregnancy. The primary outcome measure was cotinine-validated tobacco abstinence at the end of pregnancy. Secondary outcomes were cotinine-validated abstinence at 3 months postpartum and self-reported significant (>50%) reduction in daily cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* current cigarette smoker (smoked >1 cigarette in the past 7 days)
* 18 years old or older
* Willing to consider altering their smoking behavior during their pregnancy

Exclusion Criteria:

* More than 26 weeks' gestation at study entry
* No telephone access
* Not planning to live in New England for 1 year
* Unable to read and speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434
Dates: Start 2001-09; Study Completion 2005-06

PRIMARY OUTCOMES:
Biochemically-validated 7-day point prevalence tobacco abstinence at end of pregnancy

SECONDARY OUTCOMES:
Biochemically-validated 7-day point prevalence tobacco abstinence at 3 months postpartum
Self-reported significant (>50%) reduction in tobacco use
Quit attempt of >24 hours duration from enrollment to end of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital; Elyse R Park, PhD, Study Director — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tufts Health Plan, Waltham, Massachusetts

REFERENCES:
- [Result] Rigotti NA, Park ER, Regan S, Chang Y, Perry K, Loudin B, Quinn V. Efficacy of telephone counseling for pregnant smokers: a randomized controlled trial. Obstet Gynecol. 2006 Jul;108(1):83-92. doi: 10.1097/01.AOG.0000218100.05601.f8. PMID 16816060
- [Derived] Park ER, Quinn VP, Chang Y, Regan S, Loudin B, Cummins S, Perry K, Rigotti NA. Recruiting pregnant smokers into a clinical trial: using a network-model managed care organization versus community-based practices. Prev Med. 2007 Mar;44(3):223-9. doi: 10.1016/j.ypmed.2006.10.008. Epub 2007 Jan 3. PMID 17204318